CLINICAL TRIAL: NCT02405455
Title: Cerclage vs Cervical Pessary in Women With Cervical Incompetence
Acronym: CEPEIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal-Infantil Vall d´Hebron Hospital (Other)
Responsible Party: Principal Investigator, Maria Goya, MD, PhD, PhD, Maternal-Infantil Vall d´Hebron Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPEIC
Record Dates: First submitted 2015-03-16; First posted 2015-04-01 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cervical Insufficiency
Keywords: cervical insufficiency; cervical cerclage; cervical pessary
MeSH Terms: conditions — Uterine Cervical Incompetence | interventions — Cerclage, Cervical

STUDY DESIGN:
Intervention Model Description: Cervical pessary vs. Cervical cerclage
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cerclage (Experimental): Cervical cerclage.
  Interventions: Procedure: Cerclage
- Cervical pessary (Experimental): Cervical pessary
  Interventions: Device: Cervical pessary

INTERVENTIONS:
Procedure: Cerclage — Surgical procedure which consists of a strong suture being inserted into and around the cervix to close it.
  Arms: Cerclage
Device: Cervical pessary — The Arabin cervical pessary, which is CE-certified for preventing spontaneous preterm birth (CE 0482 / EN ISO 13485: 2003 annex III of the council directive 93/42 EEC). It is a vaginal device which is used to treat pregnant women for preventing spontaneous preterm birth. This device can be easily placed around the uterine cervix without pain.
  Arms: Cervical pessary

SUMMARY:
Cervical insufficiency (CI), responsible for 8% of preterm births (PB), is used to describe painless cervical dilation leading to recurrent second-trimester pregnancy losses/births of otherwise normal pregnancies. Structural weakness of cervical tissue was thought to cause or contribute to these adverse outcomes. The term has also been applied to women with one or two such losses/births or at risk for second-trimester pregnancy loss/birth. Cervical pessary and cervical cerclage are both considered as preventive treatments in women at risk for PB. This study aims to demonstrate that the cervical pessary could reduce the preterm birth rate before 37 weeks of gestation in women with prior PB due to cervical insufficiency or in women with prior PB and a short cervix in the current pregnancy.

DETAILED DESCRIPTION:
Methods/Design: This is an open-label, pilot, multicentre, prospective, randomised controlled trial (RCT). Enrolees are women with singleton pregnancies and previous PB based on CI (primary intervention, <16 weeks) or in case of previous PB and a short cervical length in current pregnancy ≤ 25 mm (secondary intervention, <24 weeks). Women are randomised (1:1) either to cervical cerclage or pessary treatment. The primary outcome is the spontaneous preterm birth rate before 34 weeks of gestation. The sample size was calculated, as a pilot study, based on the estimated population that we will be able to recruit during the duration of the trial: 60 women, 30 for each group (cervical cerclage and cervical pessary group) to observe, at least a reduction in the PB rate < 34 weeks from 34% to 27% in the pessary group, as does cerclage.

Discussion: The outcome of this study will show the effectiveness of a cervical cerclage and of a cervical pessary in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Minimum age: 18 years
* Previous PB based on CI (primary intervention, <16 weeks) or in case of previous PB and a short cervical length in current pregnancy ≤ 25 mm (secondary intervention, <24 weeks). Women are randomised (1:1) either to cervical cerclage or pessary treatment.

Exclusion Criteria:

* Major fetal abnormalities (requiring surgery or leading to infant death or severe handicap)
* Threatened preterm labour at time of randomization
* Spontaneous rupture of membranes at time of randomization
* Chorioamnionitis at time of randomization
* Active vaginal bleeding
* Placenta previa

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Spontaneous delivery before 34 complete weeks | Before 34 weeks of gestation
  Spontaneous delivery before 34 complete weeks

SECONDARY OUTCOMES:
Spontaneous delivery before 28 complete weeks | Before 28 weeks of gestation
  Spontaneous delivery before 28 complete weeks
Spontaneous delivery before 37 complete weeks | Before 37 weeks of gestation
  Spontaneous delivery before 37 complete weeks
Foetal and neonatal death | During pregnancy and during the first 28 days of newborn or NICU stay
  Foetal and neonatal death
Neonatal morbidity | 28 days of newborn or during NICU stay
  Neonatal morbidity
Maternal side effects | During pregnancy
  Maternal side effects
Maternal morbidity | during pregnancy
  Maternal morbidity
Number of participants with chorioamnionitis infection | During pregnancy
  Number of participants with chorioamnionitis infection
Hospitalisation for threatened preterm labour | During pregnancy
  Hospitalisation for threatened preterm labour

CONTACTS AND LOCATIONS:
Overall Officials: Maria Goya, PhD, Principal Investigator — Hospital Vall d'Hebrón; Andrea Gascón, MD, Principal Investigator — Hospital Vall d'Hebrón
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain